CLINICAL TRIAL: NCT05367206
Title: Department of Radiation, Sun Yat-sen University
Brief Title: Neoadjuvant Chemotherapy Followed by Chemoradiation Versus Chemoradiation for Stage IIIC Cervical Cancer Patients: A Randomized Phase III Trial
Acronym: N6C
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Junyun, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SunYat-sen University
Record Dates: First submitted 2022-05-01; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Cervical Cancer; Neoadjuvant Chemotherapy; Bulky Neoplasm
Keywords: cervical cancer; neoadjuvant chemotherapy; bulky neoplasm
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Albumin-Bound Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NAC plus RCT (Experimental): two circles of NAC with albumin-bound paclitaxel and carboplatin followed by standard chemoradiation with weekly cisplatin plus pelvic radiation
  Interventions: Drug: Albumin-Bound Paclitaxel; Drug: Carboplatin
- RCT (No Intervention): standard chemoradiation with weekly cispatin plus pelvic radiation

INTERVENTIONS:
Drug: Albumin-Bound Paclitaxel — 260mg/m2 q3w *2 circles
  Arms: NAC plus RCT
Drug: Carboplatin — AUC 5-6 q3w * 2 circles
  Arms: NAC plus RCT

SUMMARY:
Evaluate the efficacy and safety of neoadjuvant chemotherapy (NAC) with albumin-bound paclitaxel and carboplatin followed by chemoradiation therapy (CRT) for stage IIIC cervical cancer patients with carcinoma >4 cm in greatest dimension and/or lymph node >2cm in short axis.

DETAILED DESCRIPTION:
in this phase III tiral , stage IIIC cervical cancer patients with carcinoma >4 cm in greatest dimension and/or lymph node >2cm in short axis will be randomly assigned to two circles of NAC with albumin-bound paclitaxel and carboplatin followed by standard CRT with weekly cisplatin plus pelvic radiotherapy or to standard CRT alone.

The primary end point was 3-year progression-free survival (PFS). Secondary end points were response rate, 3-year locoregional control, 3-year overall survival (OS), safety, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. pathologically comfirmed : squamous cell, adenocarcinoma, or adenosquamous carcinoma of the uterine cervix；
2. FIGO (2018 International Federation of Gynecology and Obstetrics) stage IIIC with carcinoma >4 cm in greatest dimension and/or lymph node >2 cm in short axis at initial diagnosis.
3. age 18 to 70 years；
4. Eastern Cooperative Oncology Group performance status 0 to 2；
5. adequate organ function.

Exclusion Criteria:

1. not at initial diagnosis; 2. with other kind of tumor.

-

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
3-year progression-free survival ratio | up to 3 years
  the time from study randomization to 3 years, the ratio for patients without disease progression nor death.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdone, China

IPD SHARING:
Plan to Share IPD: No